CLINICAL TRIAL: NCT05478577
Title: Clinical Features and Rehabilitation Effect for Upper Limb Recovery in Patients With Stroke: Retrospective Study
Brief Title: Clinical Features and Rehabilitation Effect in Patients With Stroke
Acronym: PCR
Status: Completed | Type: Observational
Sponsor: IRCCS San Camillo, Venezia, Italy (Other)
Responsible Party: Principal Investigator, Silvia Salvalaggio, Principal Investigator, IRCCS San Camillo, Venezia, Italy
Other Study IDs: PCR 2021.20
Record Dates: First submitted 2022-07-26; First posted 2022-07-28 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Stroke
Keywords: rehabilitation; upper limb; cognitive functions; motor function
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Motor rehabilitation — Treatments for upper limb recovery (e.g. occupational therapy, technology devices, conventional therapy)

SUMMARY:
Dosage of rehabilitation therapy is a key factor in promoting motor functional recovery after stroke. To date, what is not yet known are the clinical features (e.g. the neurological profile, clinical history, motor, language and cognitive abilities), which allow the clinician to predict the recovery potential of a patient before rehabilitation, based on both the initial assessment and the various treatment pathways available in the National Health System. For these reasons, the study aims to explore clinical features and potential effect of rehabilitation dose that could influence upper limb motor recovery

DETAILED DESCRIPTION:
Dosage of rehabilitation therapy is a key factor in promoting motor functional recovery after stroke. Moreover, even though recent evidence has shown that cognitive abilities may support motor recovery, the relationship between cognitive-linguistic and motor skills in stroke patients is still a matter of research. Regarding the dose of intervention, in trials in which patients underwent 6 hours of rehabilitation per day, functional improvements in the upper limb reached clinically relevant levels, up to a difference of 8-11 points on the Fugl-Meyer Upper Extremity. To date, evidence of clinical (e.g. motor, cognitive-linguistic and neurological) and rehabilitation features that may influence upper limb recovery are still missing. Therefore, this study aims to retrospectively explore whether there is a relationship between clinical features and upper limb recovery after rehabilitation in stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* first-ever unilateral cortical-subcortical stroke, (ischemic or haemorrhagic)
* completed at least 4 weeks of rehabilitation
* preserved ability or possibility to provide informed consent.

Exclusion Criteria:

* cerebellar or bilateral stroke
* unstable medical conditions;
* diagnosis of other neurological and/or psychiatric diseases in addition to stroke;
* traumatic brain injury;
* not released informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with stroke hospitalised at San Camillo Hospital for a period of neurological rehabilitation
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment Upper Extremity | change from baseline up to 8 weeks
  Fugl-Meyer Assessment Upper Extremity is a stroke-specific scale which assesses the upper limb motor functioning in patients with post-stroke hemiplegia. There are 3 values: 0 (severe impairment), 1 (moderate impairment), 2 (preserved function). The minimum value is 0 points, which corresponds to upper limb hemiplegia. The maximum value is 66 points, which corresponds to normal motor performance.

SECONDARY OUTCOMES:
Oxford Cognitive Screen | at baseline
  Oxford Cognitive Screen is a multidomains screening tool for the assessment of cognitive functions (e.g. attention, executive functions, linguistic functions, memory). For each domain, cut-off scores are calculated according to age and education levels. There is not an overall score, but for each domain pathological performances are identified according to normative data.
Reaching Performance Scale | Change from baseline up to 8 weeks.
  Reaching Performance Scale assesses the ability of subjects to reach an object (a cone). The cone is placed at both 4-cm (close) and 30-cm (far) distance from the subject. The subject is asked to reach and grab the cone if possible. The observer evaluates the quality of reaching instead of the grip strength. The minimum value is 0 points, which corresponds to incapacity of any ability of reaching an object. The maximum value is 36 points, which corresponds to the preservation of the ability of reaching an object.
Box & Blocks Test | Change from baseline up to 8 weeks.
  The patient has to carry as much cubes as possible, one by one, from a container to another one in one minute. The test is performed with both hands.
Modified Ashworth Scale | Change from baseline up to 8 weeks.
  Spasticity is measured using the Modified Ashworth Scale of biceps muscle (Total score = 20 points). The therapist evaluates the spasticity of the muscle. There are 5 values: 0 (no increase in muscle tone), 1 (slight increase in muscle tone), 2 (more marked increase in muscle tone), 3 (considerable increase in muscle tone), 4 (affected part rigid in flexion or extension).
Functional Independence Measure | Change from baseline up to 8 weeks.
  Functional Independence Measure scale is an 18-item scale that assesses the degree of independence in carrying out activities of daily living. There are 7 values: 1 (Total Assistance or not Testable), 2 (Maximal Assistance), 3 (Moderate Assistance), 4 (Minimal Assistance), 5 (Supervision), 6 (Modified Independence), 7 (Complete Independence). The minimum values is 18 points, which corresponds to the lower level of independence in activities of daily living. The maximum value is 126 points, which corresponds to the maximum level of independence in activities of daily living.
Dose of therapy | hospitalisation period (8 weeks)
  Amount (in hours) of rehabilitation that patients underwent during hospitalisation

CONTACTS AND LOCATIONS:
Locations (1):
- San Camillo IRCCS Hospital, Venezia, Venice, Italy

IPD SHARING:
Plan to Share IPD: No